CLINICAL TRIAL: NCT06025032
Title: An Open-label, Multiple-cohort, Dose-finding, Investigator-initiated Trial to Evaluate the Safety, Tolerability, and Efficacy of HG205 RNA Base-Editing Therapy in Subjects With OTOF-p.Q829X Mutation-associated Hearing Loss
Brief Title: a Study in Subjects With Otoferlin Mutation-related Hearing Loss Using RNA Base-eDiting Therapy(SOUND)
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Huidagene stopped this program as lack of patients in China
Sponsor: HuidaGene Therapeutics Co., Ltd. (Industry)
Collaborators: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HG20501
Record Dates: First submitted 2023-08-21; First posted 2023-09-06 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Congenital Hearing Loss
Keywords: Congenital hearing loss; OTOF; Q829X; HG205; CRISPR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HG205 (Experimental): Method of Administration: Once Unilateral intracochlear injection/subject; The duration of the study for each subject includes a screening period, enrollment visit, treatment visit, a 26-week follow-up period, and a 5-year long-term safety follow-up after the injection
  Interventions: Genetic: HG205

INTERVENTIONS:
Genetic: HG205 — The study will enroll up to 2 cohorts, evaluating a starting dose plus a higher or lower dose

SUMMARY:
The purpose of the study is to determine whether HG205 as CRISPR/Cas13 RNA base-editing therapy is safe and effective for the treatment of hearing loss caused by p.Q829X mutation in OTOF gene.

ELIGIBILITY:
Inclusion Criteria:

* Male or females between 1 and 16 years of age at the time the subject/parent/legal guardian signs the informed consent form.
* Willing to adhere to the protocol as evidenced by written informed consent or parental permission and subject assent.
* Molecular diagnosis of biallelic mutations in the OTOF gene with at least one mutation being p.Q829X through collected blood samples at screening;
* Based on auditory brainstem response (ABR), clinically diagnosed sensorineural hearing loss (SNHL) with the following hearing thresholds: severe (65 dB ≤ hearing threshold < 80 dB) or profound (80 dB ≤ hearing threshold < 95 dB) or complete (hearing threshold ≥ 95 dB) hearing loss in both ears.
* Acceptable hematology, clinical chemistry, and urine laboratory parameters.

Exclusion Criteria:

* Pre-existing other hearing-loss conditions that would preclude the planned surgery or interfere with the interpretation of study endpoints or complications of surgery.
* Presence of cochlear implants in the study ear.
* Complicating systemic diseases or clinically significant abnormal baseline laboratory values.
* Complicating systemic diseases would include those in which the disease itself, or the treatment for the disease, can alter hearing function.
* Prior participation in clinical study with an investigational drug within the past six months.
* Prior gene therapy treatments.
* Any condition which leads the investigator to believe that the participant cannot comply with the protocol requirements or that may place the participant at an unacceptable risk for participation.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Incidence of otological and systemic adverse events | 26 weeks
  Number of AE(Adverse events),SAE(Serious Adverse Events),DLT(Dose Limiting Toxicities)

SECONDARY OUTCOMES:
Change from baseline in ABR(Auditory Brainstem Response) intensity threshold (decibels normal hearing level [dB nHL]) | 26 weeks
  ABR intensity threshold (decibels normal hearing level [dB nHL]) measurement
Change from baseline in hearing performance by behavioral audiometry with pure-tone audiometry | 26 weeks
  Behavioral audiometry and pure-tone audiometry measurement

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — HuidaGene Therapeutics Co., Ltd.
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No